CLINICAL TRIAL: NCT05368870
Title: Refractive Outcomes After Scleral Fixation of the Carlevale Intraocular Lens: Retrospective Study of Power Calculation Accuracy.
Brief Title: Accuracy of Intra Ocular Lens CARLEVALE Calculation
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Observational retrospective
Record Dates: First submitted 2022-04-10; First posted 2022-05-10 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Lens Diseases
MeSH Terms: conditions — Lens Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carlevale implantation
  Interventions: Procedure: Carlevale implantation

INTERVENTIONS:
Procedure: Carlevale implantation — Vitrectomy and Carlevale implantation

SUMMARY:
The purpose of this study is to assess the accuracy of intra ocular lens power calculation using the new Carlevale sutureless scleral fixation posterior chamber intra ocular lens.

DETAILED DESCRIPTION:
Retrospective comparison of refractive spherical equivalent predicted before surgery and measured after surgery in patient who underwent implantation of an sutureless scleral fixation posterior chamber intra ocular lens between October 2019 and Avril 2022 in the ophthalmology department of Poitiers Hospital and La Rochelle Hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent implantation of Carlevale between Octobre 2019 and Avril 2022 in the ophtalmologie department of Poitiers hospital and La Rochelle hospital

Exclusion Criteria:

* Post surgery best corrected visual acuity worse than 20/40
* Keratoconus
* Macular oedema

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent implantation of Carlevale between Octobre 2019 and Avril 2022 in the ophtalmologie department of Poitiers hospital and La Rochelle hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Prediction error | Between Month 1 and Month 6
  Difference between the measured and predicted post-operative refractive spherical equivalent for the intra oculaire lens power implanted

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire, Poitiers, Vienne, France

IPD SHARING:
Plan to Share IPD: Yes
Refractive data
Supporting Information: Study Protocol
Time Frame: 6 months after publication